CLINICAL TRIAL: NCT05769608
Title: A Randomized, Double-Blind, Placebo Controlled, Parallel Arm, Multicenter, Phase 2 Study to Evaluate the Efficacy and Safety of Lorundrostat in Subjects With Uncontrolled Hypertension on a Standardized Medication Regimen
Brief Title: A Pivotal Study to Evaluate the Efficacy of Lorundrostat in Subjects With Uncontrolled Hypertension on a Standardized Antihypertensive Medication Regimen
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mineralys Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MLS-101-202
Record Dates: First submitted 2023-02-24; First posted 2023-03-15 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Hypertension
Keywords: Blood pressure; Uncontrolled hypertension; Hypertension; Hypertensive; Resistant hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Placebo (Placebo Comparator): Placebo once daily for 12 weeks
  Interventions: Drug: Placebo
- Dose 1 (Experimental): lorundrostat Dose 1 once daily for 12 weeks
  Interventions: Drug: lorundrostat Dose 1
- Dose 2 (Experimental): lorundrostat Dose 1 once daily for 4 weeks then lorundrostat Dose 2 once daily for 8 weeks
  Interventions: Drug: lorundrostat Dose 2

INTERVENTIONS:
Drug: Placebo — Placebo once daily for 12 weeks
  Arms: Placebo
Drug: lorundrostat Dose 1 — lorundrostat Dose 1 once daily for 12 weeks
  Arms: Dose 1
Drug: lorundrostat Dose 2 — lorundrostat Dose 1 once daily for 4 weeks then lorundrostat Dose 2 once daily for 8 weeks for subjects who meet prespecified criteria
  Arms: Dose 2

SUMMARY:
A Phase 2 trial to evaluate the blood pressure-lowering effect of lorundrostat an aldosterone synthase inhibitor (ASI), administered as an add-on to a standardized anti-hypertensive (AHT) medication regimen, in subjects with hypertension.

DETAILED DESCRIPTION:
This study is a Phase 2 trial to evaluate the blood pressure-lowering effects of lorundrostat (an ASI), administered as add-on to a standardized anti-hypertensive (AHT) medication regimen, in subjects with hypertension.

The study consists of a standardized AHT regimen run-in period followed by a randomized, double-blind, placebo-controlled, parallel arm period. Following the double-blind period subjects may be offered the opportunity to participate in an open-label extension (OLE) study. Subjects electing to not participate in the OLE will undergo an end of study (EoS) visit approximately 2 weeks after the last dose of study drug to complete their participation in the study.

ELIGIBILITY:
Inclusion Criteria:

1. At least 18 years of age at the time of signing the informed consent form
2. At Screening: AOBP SBP of 140-180 mmHg and AOBP DBP of 65-110 mmHg, or AOBP DBP of 90-110 mmHg
3. 24-hour average ABPM SBP of 130-180 mmHg or 24-hour average ABPM DBP >80 mmHg
4. Taking between 2 and 5 AHT medications, inclusive, at Screening visit.
5. BMI of 18-40 kg/m2 inclusive at Screening

Exclusion Criteria:

1. eGFR <45 mL/min/1.73 m2 at Screening, calculated using the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) formula
2. Serum potassium >5.0 mmol/L at Screening or >4.8 mmol/L at Randomization
3. Serum sodium <135 mmol/L at Screening
4. History of heart failure, myocardial infarction, stroke, or transient ischemic attack within 6 months prior to Screening.
5. Diabetes mellitus with a glycosylated hemoglobin (HbA1c) >9% (>74.9 mmol/mol) at Screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 285 (Actual)
Dates: Start 2023-03-13 (Actual); Primary Completion 2025-01-15 (Actual); Study Completion 2025-01-15 (Actual)

PRIMARY OUTCOMES:
Change in 24-hour average ambulatory blood pressure monitoring (ABPM) systolic blood pressure (SBP) | Baseline (Randomization) to Week 12

SECONDARY OUTCOMES:
Change from baseline in 24-hour average ABPM SBP at Week 4 in subjects randomized to lorundrostat 50 mg QD compared to subjects randomized to placebo | Baseline to Week 4
Proportion of subjects with 24-hour average ABPM SBP <125 mmHg at Week 4 in subjects randomized to lorundrostat 50 mg QD compared to subjects randomized to placebo | at Week 4
Change from baseline in 24-hour average ABPM SBP at Week 4 by obesity status in subjects randomized to lorundrostat 50 mg QD compared to subjects randomized to placebo | Baseline to Week 4
Change from baseline in automated office BP (AOBP) SBP at Week 12 in subjects who were escalated to lorundrostat 100 mg QD at Week 4 (within-subjects analysis) | Baseline to Week 12
Change from baseline in 24-hour average ABPM SBP at Week 4, by number of AHT medications in the standardized AHT regimen (2 and 3) in subjects randomized to lorundrostat 50 mg QD compared to subjects randomized to placebo | Baseline to Week 4
Proportion of subjects with 24-hour average ABPM SBP <125 mmHg at Week 12 in subjects randomized to lorundrostat (by arm and pooled dosages) compared to subjects randomized to placebo | Baseline to Week 12
Change from baseline in 24-hour average ABPM SBP at Week 12 by obesity status in subjects randomized to lorundrostat (by arm and pooled dosages) compared to subjects randomized to placebo | Baseline to Week 12
Change from baseline in daytime average ABPM SBP at Week 4 and Week 12 in subjects randomized to lorundrostat 50 mg (Week 4) and by arm and pooled dosages (Week 12) compared to subjects randomized to placebo | Baseline to Week 4 and Week 12
Change from baseline in AOBP SBP at Week 4 and Week 12 in subjects randomized to lorundrostat 50 mg QD (Week 4) and by arm and pooled dosages (Week 12) compared to subjects randomized to placebo | Baseline to Week 4 and Week 12
Change from baseline in nighttime average ABPM SBP at Week 4 and Week 12 in subjects randomized to lorundrostat 50 mg QD (Week 4) and by arm and pooled dosages (Week 12) compared to subjects randomized to placebo | Baseline to Week 4 and Week 12
Change from baseline in 24-hour average ABPM SBP at Week 12, in subjects randomized to lorundrostat (pooled dosages) compared to subjects randomized to placebo | Baseline to Week 12

CONTACTS AND LOCATIONS:
Locations (104):
- United States (104):
  - Cardiology, P.C. - Birmingham, Birmingham, Alabama
  - University of Alabama at Birmingham (UAB) - Vascular Biology and Hypertension Program, Birmingham, Alabama
  - Chandler Clinical Trials, Chandler, Arizona
  - Brown Road Family Medicine, Mesa, Arizona
  - Scottsdale Clinical Trials (Elite Clinical Network), Scottsdale, Arizona
  - Fiel Family & Sports Medicine, Tempe, Arizona
  - Noble Clinical Research, Tucson, Arizona
  - Del Sol Research Management, LLC, Tucson, Arizona
  - The Medical Research Group Inc., Fresno, California
  - Marvel Clinical Research, Huntington Beach, California
  - University of California San Diego (UCSD) - Altman Clinical and Translational Research Institute (ACTRI), La Jolla, California
  - Clinical Trials Research, Lincoln, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Catalina Research Institute, Montclair, California
  - Northridge Clinical Trials, Northridge, California
  - University of California Irvine Medical Center, Orange, California
  - Triwest Research Associates, San Diego, California
  - San Jose Clinical Trials, San Jose, California
  - Blue Coast Research Center, Vista, California
  - Accelerated Enrollment Solutions (AES)- Vista, Vista, California
  - Delta Waves, Inc., Colorado Springs, Colorado
  - CMR of Greater New Haven, Hamden, Connecticut
  - Indago Research & Health Center, Inc., Hialeah, Florida
  - Clinical Neuroscience Solutions, Inc (Jacksonville), Jacksonville, Florida
  - Reserka, LLC, Miami, Florida
  - Nuovida Research Center Corp, Miami, Florida
  - Clinical Neuroscience Solutions, INC., Orlando, Florida
  - Patron Medical - Andres Patron D.O. (Patron Ventures, LLC), Pembroke, Florida
  - Progressive Medical Research, Port Orange, Florida
  - Clinical Research of West Florida, Inc., Tampa, Florida
  - The Pierone Research Institute (Elligo Health Research), Vero Beach, Florida
  - Nephrology Associates, PC - Downtown Augusta, Augusta, Georgia
  - Accel Research Sites, Decatur, Georgia
  - Georgia Clinical Research, LLC, Lawrenceville, Georgia
  - Randomize Now, Peachtree City, Georgia
  - Alta Pharmaceutical Research Center, Peachtree Corners, Georgia
  - Fellows Research Alliance, Inc, Savannah, Georgia
  - Eagle Clinical Research, Chicago, Illinois
  - The University of Chicago Medicine, Chicago, Illinois
  - GenHarp Clinical Solutions, Evergreen Park, Illinois
  - Southern Illinois School of Medicine, Springfield, Illinois
  - Franciscan Physician Network-Indiana Heart Physicians, Indianapolis, Indiana
  - Indiana Clinical Research, Merrillville, Indiana
  - The Research Group of Lexington, LLC, Lexington, Kentucky
  - Advanced Internal Medicine, PLLC (Elligo Health Research), Paducah, Kentucky
  - Versailles Family Medicine, Versailles, Kentucky
  - Cambridge Clinical Trials, Alexandria, Louisiana
  - Pennington Biomedical Research Center, Baton Rouge, Louisiana
  - Boston Clinical Trials, Boston, Massachusetts
  - ActivMed Practices & Research, LLC, Methuen, Massachusetts
  - Saint Louis University, St Louis, Missouri
  - Quality Clinical Research Inc. (QCR) - Omaha, Omaha, Nebraska
  - Henderson Clinical Trials, Henderson, Nevada
  - Las Vegas Clinical Trials, Las Vegas, Nevada
  - Oasis Clinical Trials, Las Vegas, Nevada
  - Renown Regional Medical Center, Reno, Nevada
  - Seacoast Kidney & Hypertension Specialist, Portsmouth, New Hampshire
  - Albany Medical College Div of Community Endocrinology, Albany, New York
  - University of Buffalo, Buffalo, New York
  - Columbia University, New York, New York
  - Marian David, MD, PC (Elligo Health Research), New York, New York
  - Triad Internal Medicine, Asheboro, North Carolina
  - Asheville Clinical Trials (Elite Clinical Network), Asheville, North Carolina
  - Duke University Medical Center Heart Center Clinical Research Unit, Durham, North Carolina
  - East Carolina University (ECU) Physicians - East Carolina Heart Institute - East Carolina University Location, Greenville, North Carolina
  - Lucas Research, Inc., New Bern, North Carolina
  - Iredell Memorial Hospital, Inc (Elligo Health Research), Statesville, North Carolina
  - Lillestol Research LLC, Fargo, North Dakota
  - Research Innovations (Elligo Health Research), Beavercreek, Ohio
  - Diabetes and Endocrinology Associates of Stark County, Inc., Canton, Ohio
  - Intrepid Research, Cincinnati, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Centricity Research (Aventiv Research) - Women's Health, Dublin, Ohio
  - STAT Research, Springboro, Ohio
  - Williamette Valley Clincial Studies, Eugene, Oregon
  - AMS Cardiology, Horsham, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Accelerated Enrollment Solutions (AES)- Anderson, Anderson, South Carolina
  - WR- Notus Clinical Trials, LLC, Charleston, South Carolina
  - Coastal Carolina Research Center, North Charleston, South Carolina
  - Chattanooga Medical Research, Chattanooga, Tennessee
  - Lifedoc Research, Memphis, Tennessee
  - Clinical Neuroscience Solutions, Inc, Memphis, Tennessee
  - Vanderbilt University Medical Center (VUMC), Nashville, Tennessee
  - Elligo Health Research, Austin, Texas
  - Punzi Medical Center, Carrollton, Texas
  - David Turbay, MD, PLLC (Elligo Health Research), El Paso, Texas
  - Houston Methodist Research Institute, Houston, Texas
  - Juno Research LLC, Houston, Texas
  - Gulf Coast Clinical Research, Houston, Texas
  - Medical Colleagues of Texas, LLP (Elligo Health Research), Katy, Texas
  - Synergy Groups Medical - Bissonet Site, Katy, Texas
  - PRX Research - Mesquite, Mesquite, Texas
  - Medical Colleagues of Texas, LLP (Elligo Health Research), Paris, Texas
  - ACRC Trials, Plano, Texas
  - Clinical Investigations of Texas (CIT), Plano, Texas
  - Sun Research Institute (SRI) - San Antonio, San Antonio, Texas
  - San Antonio Clinical Trials, San Antonio, Texas
  - Sugar Lakes Family Practice (Elligo Health Research), Sugar Land, Texas
  - The University of Utah, Salt Lake City, Utah
  - Burke Internal Medicine, Burke, Virginia
  - Charlottesville Medical Research, Charlottesville, Virginia
  - Eastern Virginia Medical School, Norfolk, Virginia
  - Centricity Research (IACT Health) (Hampton Roads Center For Clinical Research, Inc.)) - Suffolk Multispecialty Research, Suffolk, Virginia

REFERENCES:
- [Derived] Laffin LJ, Kopjar B, Melgaard C, Wolski K, Ibbitson J, Bhikam S, Weir MR, Ofili EO, Mehra R, Luther JM, Cohen DL, Sarraju A, Wilkinson MJ, Flack JM, Rodman D, Nissen SE; Advance-HTN Investigators. Lorundrostat Efficacy and Safety in Patients with Uncontrolled Hypertension. N Engl J Med. 2025 May 8;392(18):1813-1823. doi: 10.1056/NEJMoa2501440. Epub 2025 Apr 23. PMID 40267417